CLINICAL TRIAL: NCT07017218
Title: The Impact of Immune Nutrition on Nutritional and Immune Status of Head and Neck Cancer Patients During Radiotherapy
Brief Title: Immunonutrition Effects on Nutrition and Immunity in HNC During Radiotherapy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: First Affiliated Hospital of Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Tao Zhang, Chief of Radiotherapy department, First Affiliated Hospital of Chongqing Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT2025-06
Record Dates: First submitted 2025-03-24; First posted 2025-06-12 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-05

CONDITIONS: Head and Neck Cancer; Nutrition
Keywords: Head and neck cancer; immunonutrition; radiation
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Immunonutrition (Experimental)
  Interventions: Dietary Supplement: IMPACT

INTERVENTIONS:
Dietary Supplement: IMPACT — immune enhanced formula enriched in arginine, n-3 PUFA and nucleotide

SUMMARY:
Head and neck cancer (HNC) is one of the most common types of malignant tumors, often leading to malnutrition due to its complex anatomical location near many functional organs. Radiotherapy, an essential treatment modality for HNC, can exacerbate malnutrition, potentially causing radiotherapy failure. Both domestic and international guidelines advocate early nutritional intervention for HNC patients at risk of malnutrition; however, specific recommendations on the type of nutritional treatment are lacking. Immunonutrition has shown promise in regulating the immune microenvironment, enhancing immune response, and reducing radiotherapy side effects compared to conventional nutritional interventions. However, there is a lack of studies focusing on immunonutritional therapy during the radiotherapy process for HNC in China. Therefore, this study aims to investigate the effects of immunonutrition on nutritional status, immune function, and quality of life (QoL) in head and neck cancer (HNC) patients undergoing radiotherapy.

This prospective interventional study enrolled 48 head and neck cancer (HNC) patients scheduled to undergo radiotherapy (with or without concurrent chemotherapy). All participants received an immunonutrition formula supplemented with arginine, ω-3 fatty acids, and nucleotides. Throughout the radiotherapy course, certified dietitians and oncology nurses provided standardized nutritional guidance based on a five-step nutritional management protocol. Primary outcomes included:Radiotherapy-related adverse events (e.g., mucositis, dysphagia) assessed at four time points during radiotherapy (weeks 1, 3, 5, and 7) using CTCAE v4.0 criteria;Longitudinal changes in nutritional status (serum albumin, BMI), immune-related biomarkers , and quality of life were assessed at baseline, mid-radiotherapy (week 4), and post-treatment (week 7).

ELIGIBILITY:
Inclusion Criteria:

* Patients must be histologically or cytologically confirmed to have head and neck cancer (HNC).
* Scheduled for radiotherapy with or without concurrent chemotherapy.
* Willingness to sign informed consent voluntarily.
* Aged between 18 and 75 years old.
* Karnofsky Performance Status (KPS) score ≥70.
* Hematological and biochemical parameters within the following ranges:
* White blood cell count (WBC) ≥3.5×10^9/L
* Hemoglobin (Hb) ≥90 g/L
* Platelet count (PLT) ≥100×10^9/L
* Serum albumin (ALB) ≥30 g/L
* Total bilirubin ≤1.5 times the upper limit of normal (ULN)
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5 - times ULN
* Life expectancy of at least 6 months.
* No severe malnutrition at baseline (e.g., body mass index [BMI] >18.5 kg/m²).

Exclusion Criteria:

* Prior history of radiation therapy or biological therapy targeting the head and neck region.
* History of other malignant tumors in the past 5 years, except for adequately treated non-melanoma skin cancer or carcinoma in situ.
* Severe systemic diseases, such as uncontrolled diabetes mellitus, severe cardiovascular disease, or chronic renal failure.
* Pregnancy or lactation.
* Drug or alcohol abuse.
* Participation in other clinical trials within the last 3 months.
* Known allergies or contraindications to the nutritional formulations used in this study.
* Mental disorders or cognitive impairments that may affect compliance with the study protocol.
* Inability to tolerate oral nutritional supplements (ONS).
* Any condition deemed by the investigator to potentially interfere with the study objectives or participant safety

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-06-20 (Estimated); Primary Completion 2025-11-30 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Severity of oral mucositis measured by CTCAE v4.0 (Grades 0-4) | Assessed weekly during radiotherapy at weeks 1, 3, 5, and 7 of treatment
  The grades of oral mucositis were measured and recorded by our professional nutritionists at four time periods during radiotherapy. The classification standard of oral mucositis was based on CTCAE v4.0 (Grade 0: asymptomatic; Grade I: Erythema appears on the oral mucosa, accompanied by pain, but it does not affect eating; Grade II: Erythema and ulcers appear on the oral mucosa, and solid food can be consumed; Grade III: Severe erythema and ulcers appear on the oral mucosa, and solid food cannot be consumed; Grade IV: Ulcers have fused into patches, with necrosis, and the patient is unable to eat)

SECONDARY OUTCOMES:
Change in body weight (kg) from baseline | at baseline, mid-radiotherapy (week 4), and post-treatment (week 7)
  Measured in kilograms using a calibrated scale, with participants in light clothing and fasting overnight
Change in Body Mass Index (BMI, kg/m²) from baseline | at baseline, mid-radiotherapy (week 4), and post-treatment (week 7)
  Calculated from measured weight and height (BMI = weight[kg] / height[m]²)
Change in serum albumin concentration (g/dL) from baseline | at baseline, mid-radiotherapy (week 4), and post-treatment (week 7)
  Measured from venous blood samples using standardized clinical laboratory assays